CLINICAL TRIAL: NCT05385575
Title: A Randomized, Double-blind and Placebo-controlled Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of KN056 in Healthy Participants
Brief Title: A Study to Evaluate Effects of KN056 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Alphamab Co., Ltd. (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: KN056-A-101
Record Dates: First submitted 2022-05-18; First posted 2022-05-23 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2023-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Cohort 1 (Experimental): Participant will receive 0.1mg of single dose by subcutaneous injection of KN056
  Interventions: Drug: KN056 (0.1mg)
- Cohort 2 (Experimental): Participant will receive 0.3mg of single dose by subcutaneous injection of KN056
  Interventions: Drug: KN056 (0.3mg)
- Cohort 3 (Experimental): Participant will receive 1.0mg of single dose by subcutaneous injection of KN056 or placebo
  Interventions: Drug: KN056 (1.0mg)
- Cohort 4 (Experimental): Participant will receive 3.0mg single subcutaneous dose of KN056 or placebo
  Interventions: Drug: KN056 (3.0mg)
- Cohort 5 (Experimental): Participant will receive 6.0mg of single dose by subcutaneous injection of KN056 or placebo
  Interventions: Drug: KN056 (6.0mg)
- Cohort 6 (Experimental): Participant will receive 12.0mg of single dose by subcutaneous injection of KN056 or placebo
  Interventions: Drug: KN056 (12.0mg)
- Cohort 7 (Experimental): Participant will receive 18.0mg of single dose by subcutaneous injection of KN056 or placebo
  Interventions: Drug: KN056 (18.0mg)

INTERVENTIONS:
Drug: KN056 (0.1mg) — The participants will receive assigned single dose of KN056 on Day 1
  Arms: Cohort 1
Drug: KN056 (0.3mg) — The participants will receive assigned single dose of KN056 on Day 1
  Arms: Cohort 2
Drug: KN056 (1.0mg) — The participants will receive assigned single dose of KN056 or placebo on Day 1
  Arms: Cohort 3
Drug: KN056 (3.0mg) — The participants will receive assigned single dose of KN056 or placebo on Day 1
  Arms: Cohort 4
Drug: KN056 (6.0mg) — The participants will receive assigned single dose of KN056 or placebo on Day 1
  Arms: Cohort 5
Drug: KN056 (12.0mg) — The participants will receive assigned single dose of KN056 or placebo on Day 1
  Arms: Cohort 6
Drug: KN056 (18.0mg) — The participants will receive assigned single dose of KN056 or placebo on Day 1
  Arms: Cohort 7

SUMMARY:
This is a Phase 1, First-in-human, double-blinded, placebo-controlled study which aims to investigate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and the immunogenicity of KN056 in healthy participants.

DETAILED DESCRIPTION:
KN056 is a biological innovative drug developed as a treatment for type 2 diabetes. It is a recombinant human Fc-fused GLP-1 variant protein. GLP-1 can activate the intracellular pathway to cause the elevation of cAMP, thereby promoting insulin secretion and inhibiting glucagon secretion.

The study will involve a single ascending (increasing) dose (SAD) study and will enroll up to 46 healthy participants across 7 dosing groups.

Cohort 1 - 0.1mg (2 participants, both receiving KN056 separated by at least 1 day) Cohort 2 - 0.3mg (4 participants, dosed as 2 +2, separated by a safety observation of at least 3 days) Cohort 3 - 1.0mg (6 participants receiving KN056 + 2 receiving placebo) Cohort 4 - 3.0mg (6 participants receiving KN056 + 2 receiving placebo) Cohort 5 - 6.0mg (6 participants receiving KN056 + 2 receiving placebo) Cohort 6 - 12.0mg (6 participants receiving KN056 + 2 receiving placebo) Cohort 7 - 18.0mg (6 participants receiving KN056 + 2 receiving placebo) In Cohort 3 to 6; the first 2 subjects will be as sentries, and will be injected with KN056 or placebo randomly: at least 3 days after 2 sentries' administration, the remaining 6 participants will be randomized to receive KN056 or placebo in a 5:1 ratio. Additional dose group: the number and randomization of Cohort 7 participants are identical to those in Cohort 3 to Cohort 6.

The dose will be given as a subcutaneous (SC) injection into the abdomen.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects (not be breastfeeding);
2. Aged between 18 and 55 (including thresholds) at the time of signing Informed Consent Form;
3. Body mass index (BMI) between 18.5 and 35.0 kg/m2 (excluding the threshold);
4. 3.5mmol/L(63 mg/dL) less than or equal to Fasting blood glucose level less than 6.1mmol/L(110 mg/dL).
5. Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures and are willing to follow study restrictions;
6. Are able and willing to sign the ICF.

Exclusion Criteria:

1. Those who have a history of chronic diseases or are currently suffering from obvious systemic diseases, such as diseases of cardiovascular system, respiratory system, endocrine and metabolic system, urinary system, digestive system, blood system, autoimmune system, neurological or psychiatric system, bacterial or viral infection;
2. History or presence of pancreatitis (history of chronic pancreatitis or idiopathic acute pancreatitis)
3. History of GI disorder (for example, relevant esophageal reflux or gall bladder disease) or any GI disease which impacts gastric emptying (for example, gastric bypass surgery, pyloric stenosis, with the exception of appendectomy) or could be aggravated by GLP-1 analogs or DPP-IV inhibitors;
4. Participants with dyslipidemia (Total Cholesterol more than 6mmol/L and/or Triglyceride more than or equal to 1.7 mmol/L);
5. Participants had cholecystolithiasis (removal of gallstones) and/or cholecystectomy (removal of gall bladder) in the past;
6. A personal or family history of medullary thyroid cancer or multiple endocrine adenoma syndrome type 2 (MEN2);
7. Allergies to GLP-1 analogues, or KN056 related compounds;
8. A history of medicine abuse/dependence or narcotics abuse within 1 year prior to the screening and/or show positive findings on urinary drug screening;
9. Previous alcoholism or have regular alcohol consumption (drinking more than 14 units of alcohol per week in the 3 months prior to the screening, are unwilling to stop alcohol consumption from at least 48 hours before landing in Phase I ward (D-2) to the end of discharge from the clinical research unit (CRU), or are unwilling to limit intake to a maximum of 2 units per day on all other days from screening through follow-up (1 unit =12oz or 360 mL of beer; 5oz or 150 mL of wine; 1.5oz or 45 mL of distilled spirits);
10. Smokers who have smoked more than 10 cigarettes or equivalent in nicotine (e-cigarettes/vaping) daily within 3 months prior to screening or are unwilling to refrain from smoking on the day of drug administration or are unable to abide by clinical research unit (CRU) restrictions;
11. Blood donation or blood loss ≥ 300 mL within 3 months prior to screening (except female physical blood loss), or blood/blood components donation planned during the trial or within 1 month after the final study visit;
12. Those who participated in any drug/vaccine clinical trial, and the last administration of the trial was within 3 months or 5 half-lives of the drug/vaccine prior to dosing of study drug, whichever is longer;
13. Received vaccination within 14 days prior to screening, or have vaccination schedule during the trial (from screening to the final visit), including inactivated vaccine, live attenuated vaccine, recombinant protein vaccine, recombinant adenovirus vaccine, RNA vaccine, DNA vaccine, COVID-19 vaccine;
14. Use medication (including prescription drugs, over-the-counter drugs, herbal medicine) with the exception of vitamin/mineral supplements, paracetamol, topical medication, and contraceptives within 14 days prior to dosing;
15. Have abnormal and clinically significant results of physical examination, vital signs, abdominal B-ultrasonography (liver, gallbladder, pancreas, spleen and kidneys) or thyroid B-ultrasonography, and may increases the risks associated with participating in the study;
16. Have abnormal and clinically significant results of Hematology, Urinalysis, blood biochemistry, serum lipase, calcitonin, thyroid function and glycosylated hemoglobin (HbA1c>40mmol/mol (5.8%)) and may increases the risks of participants in the study;
17. ECG shows increased heart rate (>100 beats/min), arrhythmia, significant QT/QTc interval prolongation (QTcF (Frederica values) >450ms for males and > 470ms for females) and other manifestations, which are clinically significant;
18. Evidence of hepatitis B or positive hepatitis B surface antigen at screening; evidence of hepatitis C or hepatitis C antibody at screening; evidence of AIDS and/or positive HIV antibodies at screening; evidence of syphilis and/or syphilis test is positive at screening;
19. The result of coronavirus nucleic acid test (COVID-19) is positive at screening or admission (Day-2)
20. Participants that refuse to stay abstinent, and refuse to consistently use a form of highly effective birth control in combination with a barrier method if heterosexually active starting at Screening (signing the ICF) and continuing throughout the clinical study period, and to 3 months after administration of KN056 or Placebo, or participants tell that their partners refuse to do so;

    Examples of highly effective forms of contraception include:
    * Implant contraceptive (e.g. Jadelle®)
    * Intra-uterine device (IUD) containing either copper or levonorgestrel (e.g. Mirena®)
    * Male sterilization (vasectomy)
    * Female sterilization (e.g. bilateral tubal ligation ('clipping or tying tubes') or hysterectomy)
    * Injectable contraceptive (e.g. Depo Provera)
    * Oral Contraceptive Pill (combined hormonal contraceptive pill or progestogen-only 'mini-pill')

    These requirements do not apply to female participants in a same sex relationship and female participants of nonchildbearing potential.

    Female participants of nonchildbearing potential should meet one of the following conditions:
    * Must have a confirmed clinical history of sterility (documented hysterectomy, bilateral salpingectomy, or bilateral oophorectomy, as confirmed by review of the subjects' medical records, medical examination, or medical history interview)
    * Must be postmenopausal as defined as: amenorrhea for ≥ 12 months prior to screening and a laboratory confirmed serum follicle-stimulating hormone (FSH) level ≥ 40 IU/L at screening.
21. Female participants of childbearing potential (no matter homosexuality or heterosexuality) with positive pregnancy test at Screening and Day -1;
22. Participants that plan to donate sperms/eggs from dosing until 3 months after administration of KN056 or Placebo;
23. Participants with any inappropriate factor for participation in this study considered by the investigator or sponsor;

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Number of treatment-emergent adverse events (TEAEs) and treatment related (TRAEs). TEAEs will be measured as per the Common Terminology Criteria for Adverse Events (CTCAE) v 5.0. | Up to 45 days
Severity of TEAEs and treatment related TEAEs. TEAEs will be measured as per the Common Terminology Criteria for (CTCAE) v5.0 | Up to 45 days
Number of participants with abnormal clinically significant laboratory results. | Up to 45 days
  Clinical laboratory includes hematology, biochemistry, lipase, calcitonin, thyroid function, Abdominal and thyroid B-ultrasonography, and urinalysis.
Number of participants with abnormal clinically significant vital signs. | Up to 45 days
  Vital signs include Includes blood pressure (systolic and diastolic), respiration, temperature and pulse.
Number of participants with abnormal clinically significant electrocardiogram (ECG) | Up to 45 days
  12-lead ECG will be performed.

SECONDARY OUTCOMES:
To evaluate the pharmacokinetic parameters of KN056. Pharmacokinetic parameters will be estimated using non-compartment model analysis with Phoenix WinNolin 8.0 | Day 1, Day 7, Day 14, Day 21, Day 28, Day 42
  Parameters: AUC0-last, AUC0-inf, MRT, Tmax, Cmax or above and T1/2, CL/F, Vz/F and so on.
Immunogenicity of KN056 | Up to 45 days
  The immunogenicity of KN056 will be evaluated by detection of ADA, and ADA titer and NAb will be detected in ADA positive samples
The efficacy of KN056 by analyzing fasting blood glucose | Up to 45 days
The efficacy of KN056 through Oral Glucose Tolerance test (OGTT) | Up to 45 days
The efficacy of KN056 by analyzing HbA1c (Glycosylated hemoglobin) changes | Up to 45 days

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Cole, Principal Investigator — New Zealand Clinical Research
Locations (1):
- Alexandra Cole, Christchurch, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No